CLINICAL TRIAL: NCT05369286
Title: A Phase 1 Study to Evaluate the Safety and Efficacy of Max-40279-01 in Combination With Toripalimab in Patients With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety and Efficacy of Max-40279 and Toripalimab in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAX-40279-008
Record Dates: First submitted 2022-04-26; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- dose level 1 of max-40279 combined dose level 1 of toripalimab (Experimental): "MAX-40279-01" and "toripalimab"
  Interventions: Drug: "MAX-40279-01" and "Toripalimab"
- dose level 2 of max-40279 combined dose level 1 of toripalimab (Experimental): "MAX-40279-01" and "toripalimab"
  Interventions: Drug: "MAX-40279-01" and "Toripalimab"
- dose level 2 of max-40279 combined dose level 2 of toripalimab (Experimental): "MAX-40279-01" and "toripalimab"
  Interventions: Drug: "MAX-40279-01" and "Toripalimab"
- dose level 3 of max-40279 combined dose level 2 of toripalimab (Experimental): "MAX-40279-01" and "toripalimab"
  Interventions: Drug: "MAX-40279-01" and "Toripalimab"
- recommend dose of max-40279 combined recommend dose level of toripalimab (Experimental): "MAX-40279-01" and "toripalimab"
  Interventions: Drug: "MAX-40279-01" and "Toripalimab"

INTERVENTIONS:
Drug: "MAX-40279-01" and "Toripalimab" — "MAX-40279-01"combined with "Toripalimab"

SUMMARY:
This include two parts, part 1 is a dose escalation study and part 2 is a dose expansion study.

DETAILED DESCRIPTION:
This study is a study of Max-40279-01 in combination with toripalimab in patients with advanced solid tumors. This study includes two Parts, the Part 1 will assess the safety and efficacy of the preset several dose levels of Max-40279-01 and toripalimab, and recommend a dose level of Max-40279-01 combined toripalimab for stage 2. The part 2 is designed to study the efficacy and safety of max-40279-01 combined toripalimab in advanced solid tumors or certain specific tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented local advanced or metastatic solid tumor.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >3 months.
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia, peripheral sensory neuropathy grade ≤ 2 and those listed in specific exclusion criteria) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0) at the time of randomization.
3. Inadequate organ or bone marrow function.
4. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
5. Pregnant or breast-feeding woman.
6. Known allergies, hypersensitivity, or intolerance to Max-40279-01 the excipients of these treatments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
DLTs | 21 days
  Dose limiting toxicity
Incidence of Treatment-Emergent Adverse Events | 24 months
  Safety and tolerability assessed by incidence and severity of adverse events

SECONDARY OUTCOMES:
Subsequent clinical recommended dose | 12 months
  Subsequent clinical recommended dose
Cmax | Approximately 6 months
  Maximum plasma drug concentration of Max-40279
Tmax | Approximately 6 months
  Time to maximum plasma concentration of Max-40279
AUC | Approximately 6 months
  Area under the time-concentration curve of Max-40279
T1/2 | Approximately 6 months
  Half-life of Max-40279
The blood concentration of toripalimab | Approximately 6 months
  The blood concentration of toripalimab
ADA | 6 months
  Anti-drug antibody of toripalimab
The efficacy end points: ORR、DCR，PFS，DOR，OS | 24 months
  Objective response rate,Disease control rate,Progression-free survival,Duration of response,Overall survival
the correlation of efficacy and the expression level and mutations of FGFR1OP2, its related proteins and inflammatory factors | 24 months
  the correlation of efficacy and the expression level and mutations of FGFR1OP2, its related proteins and inflammatory factors

CONTACTS AND LOCATIONS:
Overall Officials: xiangen MD Lu, Ph.D, Study Chair — Institute of The Sixth Affiliated Hospital Sun Yat-sen University
Locations (1):
- Institute of The Sixth Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No